CLINICAL TRIAL: NCT00986817
Title: Efficacy of Terlipressin in Cirrhotic Patients With Recidivation Ascites Treated With Paracentesis and Albumin. A Multi-center Randomized Controlled Study
Brief Title: Terlipressin in Cirrhotic Patients With Recidivation Ascites Treated With Paracentesis and Albumin
Acronym: TERAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P071215
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Cirrhosis
Keywords: Refractory ascites; Cirrhosis Terlipressin; Paracentesis
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Terlipressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terlipressin (Experimental)
  Interventions: Drug: Terlipressin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Terlipressin — Albumin perfusions at the dose 8 g/l of removed ascites and Terlipressin (1mg), administrated before and at the end of the paracentesis.
  Arms: Terlipressin
Drug: Placebo — albumin perfusion at the dose 8 g/l of removed ascites and placebo, administrated before and at the end of the paracentesis.
  Arms: Placebo

SUMMARY:
Ascites is a common complication of cirrhosis. Sodium restriction and diuretics are the first step treatment. Refractory ascites (not responding to first step treatment) is treated with repeated large volume paracentesis followed by intra venous albumin expansion. In pilot studies vasoconstrictor agents such as terlipressin have shown beneficial effect on ascites production. Therefore the investigators will study the effect of combined therapy with albumin and terlipressin on recidivation ascites.

DETAILED DESCRIPTION:
About 30% of cirrhotic patients will develop ascites. Sodium restriction and diuretics are the first step treatment. Total paracentesis is used in patients with cirrhosis and tense ascites. Paracentesis alone was found to induce a decrease in effective arterial blood volume. This circulatory dysfunction may induce inhospital complications such as impaired renal function or hyponatremia and is associated with a significant reduction in long term survival. Intravenous albumin administration after paracentesis has been shown to prevent the post paracentesis decrease in arterial blood volume. Paracentesis also induces arteriolar vasodilation which plays a major role in initiating the decrease in arterial blood volume. Therefore, administration of a vasoconstrictor may decrease paracentesis induced arteriolar vasodilation and prevent the resulting decrease in effective arterial blood volume. Two randomised pilot studies suggest that Terlipressin may be as effective as intravenous albumin in preventing a decrease in effective arterial blood volume in patients with cirrhosis treated by paracentesis for tense ascites. The combined treatment, albumin plus terlipressin, could have additional effect and may improve ascites in such patients. In several studies the combined therapy, albumin plus terlipressin, has shown beneficial effect in cirrhotic patients with hepatorenal syndrome characterized by a sever decrease in arterial blood volume and vasodilation. In these studies, combined therapy was well tolerated.The aim of this study is to compare ascites relapse between two groups of cirrhotic patients with recidivation ascites treated by paracentesis and intravenous albumin perfusion plus terlipressin or placebo. In this double blind randomized multi-center trial, all patients receive albumin perfusion at the dose 8 g/l of removed ascites and Terlipressin (1mg) or placebo, administrated before and at the end of the paracentesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years old and more with cirrhosis and refractory ascites define by the international ascites club.
* Vital status non engaged in the 2 months

Exclusion Criteria:

* cardiovascular disease : previous or actual angina pectoralis, myocardial infarction, heart failure, rhythm or conduction disorders, repolarisation abnormality on ECG
* respiratory disease: previous or actual chronic pulmonary insufficiency, asthma
* uncontrolled hypertension
* acute portal vein thrombosis (less then 3 months) or currently treated.
* chronic renal insufficiency (creatin > 15 mg/L)
* severe hepatic encephalopathy
* Alcoholic hepatitis or gastrointestinal bleeding in the last 3 months
* hepatocellular carcinoma
* severe illness with life threatening
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-11; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Mean number of paracentesis between the 2 groups over a 6 months period | 6 months

SECONDARY OUTCOMES:
Total ascites retrieval | 6 months
Number of cirrhosis complications groups | 6 months
Liver transplantation and deaths | 6 months
Terlipressin safety | 6 months
Mean number of days of hospitalization | 6 months
Delay between inclusion and the first rehospitalisation for ascites retrieval | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Carbonell, MD, Principal Investigator — Hôpital Saint Antoine
Locations (1):
- CARBONELL Nicolas, Paris, Paris, France

REFERENCES:
- [Background] Runyon BA. Management of adult patients with ascites caused by cirrhosis. Hepatology. 1998 Jan;27(1):264-72. doi: 10.1002/hep.510270139. PMID 9425946
- [Background] Gines P, Quintero E, Arroyo V, Teres J, Bruguera M, Rimola A, Caballeria J, Rodes J, Rozman C. Compensated cirrhosis: natural history and prognostic factors. Hepatology. 1987 Jan-Feb;7(1):122-8. doi: 10.1002/hep.1840070124. PMID 3804191
- [Background] Moore KP, Wong F, Gines P, Bernardi M, Ochs A, Salerno F, Angeli P, Porayko M, Moreau R, Garcia-Tsao G, Jimenez W, Planas R, Arroyo V. The management of ascites in cirrhosis: report on the consensus conference of the International Ascites Club. Hepatology. 2003 Jul;38(1):258-66. doi: 10.1053/jhep.2003.50315. PMID 12830009
- [Background] Gines A, Fernandez-Esparrach G, Monescillo A, Vila C, Domenech E, Abecasis R, Angeli P, Ruiz-Del-Arbol L, Planas R, Sola R, Gines P, Terg R, Inglada L, Vaque P, Salerno F, Vargas V, Clemente G, Quer JC, Jimenez W, Arroyo V, Rodes J. Randomized trial comparing albumin, dextran 70, and polygeline in cirrhotic patients with ascites treated by paracentesis. Gastroenterology. 1996 Oct;111(4):1002-10. doi: 10.1016/s0016-5085(96)70068-9. PMID 8831595
- [Background] Ruiz-del-Arbol L, Monescillo A, Jimenez W, Garcia-Plaza A, Arroyo V, Rodes J. Paracentesis-induced circulatory dysfunction: mechanism and effect on hepatic hemodynamics in cirrhosis. Gastroenterology. 1997 Aug;113(2):579-86. doi: 10.1053/gast.1997.v113.pm9247479.
- [Background] Gines P, Tito L, Arroyo V, Planas R, Panes J, Viver J, Torres M, Humbert P, Rimola A, Llach J, et al. Randomized comparative study of therapeutic paracentesis with and without intravenous albumin in cirrhosis. Gastroenterology. 1988 Jun;94(6):1493-502. doi: 10.1016/0016-5085(88)90691-9. PMID 3360270
- [Background] Moreau R, Lebrec D. The use of vasoconstrictors in patients with cirrhosis: type 1 HRS and beyond. Hepatology. 2006 Mar;43(3):385-94. doi: 10.1002/hep.21094. PMID 16496352
- [Background] Moreau R, Valla DC, Durand-Zaleski I, Bronowicki JP, Durand F, Chaput JC, Dadamessi I, Silvain C, Bonny C, Oberti F, Gournay J, Lebrec D, Grouin JM, Guemas E, Golly D, Padrazzi B, Tellier Z. Comparison of outcome in patients with cirrhosis and ascites following treatment with albumin or a synthetic colloid: a randomised controlled pilot trail. Liver Int. 2006 Feb;26(1):46-54. doi: 10.1111/j.1478-3231.2005.01188.x. PMID 16420509
- [Background] Moreau R, Asselah T, Condat B, de Kerguenec C, Pessione F, Bernard B, Poynard T, Binn M, Grange JD, Valla D, Lebrec D. Comparison of the effect of terlipressin and albumin on arterial blood volume in patients with cirrhosis and tense ascites treated by paracentesis: a randomised pilot study. Gut. 2002 Jan;50(1):90-4. doi: 10.1136/gut.50.1.90. PMID 11772973
- [Background] Singh V, Kumar R, Nain CK, Singh B, Sharma AK. Terlipressin versus albumin in paracentesis-induced circulatory dysfunction in cirrhosis: a randomized study. J Gastroenterol Hepatol. 2006 Jan;21(1 Pt 2):303-7. doi: 10.1111/j.1440-1746.2006.04182.x. PMID 16460491
- [Background] Solanki P, Chawla A, Garg R, Gupta R, Jain M, Sarin SK. Beneficial effects of terlipressin in hepatorenal syndrome: a prospective, randomized placebo-controlled clinical trial. J Gastroenterol Hepatol. 2003 Feb;18(2):152-6. doi: 10.1046/j.1440-1746.2003.02934.x. PMID 12542598
- [Background] Ortega R, Gines P, Uriz J, Cardenas A, Calahorra B, De Las Heras D, Guevara M, Bataller R, Jimenez W, Arroyo V, Rodes J. Terlipressin therapy with and without albumin for patients with hepatorenal syndrome: results of a prospective, nonrandomized study. Hepatology. 2002 Oct;36(4 Pt 1):941-8. doi: 10.1053/jhep.2002.35819. PMID 12297842
- [Background] Moreau R, Durand F, Poynard T, Duhamel C, Cervoni JP, Ichai P, Abergel A, Halimi C, Pauwels M, Bronowicki JP, Giostra E, Fleurot C, Gurnot D, Nouel O, Renard P, Rivoal M, Blanc P, Coumaros D, Ducloux S, Levy S, Pariente A, Perarnau JM, Roche J, Scribe-Outtas M, Valla D, Bernard B, Samuel D, Butel J, Hadengue A, Platek A, Lebrec D, Cadranel JF. Terlipressin in patients with cirrhosis and type 1 hepatorenal syndrome: a retrospective multicenter study. Gastroenterology. 2002 Apr;122(4):923-30. doi: 10.1053/gast.2002.32364. PMID 11910344
- [Background] Halimi C, Bonnard P, Bernard B, Mathurin P, Mofredj A, di Martino V, Demontis R, Henry-Biabaud E, Fievet P, Opolon P, Poynard T, Cadranel JF. Effect of terlipressin (Glypressin) on hepatorenal syndrome in cirrhotic patients: results of a multicentre pilot study. Eur J Gastroenterol Hepatol. 2002 Feb;14(2):153-8. doi: 10.1097/00042737-200202000-00009. PMID 11981339
- [Background] Uriz J, Gines P, Cardenas A, Sort P, Jimenez W, Salmeron JM, Bataller R, Mas A, Navasa M, Arroyo V, Rodes J. Terlipressin plus albumin infusion: an effective and safe therapy of hepatorenal syndrome. J Hepatol. 2000 Jul;33(1):43-8. doi: 10.1016/s0168-8278(00)80158-0. PMID 10905585
- [Background] Mulkay JP, Louis H, Donckier V, Bourgeois N, Adler M, Deviere J, Le Moine O. Long-term terlipressin administration improves renal function in cirrhotic patients with type 1 hepatorenal syndrome: a pilot study. Acta Gastroenterol Belg. 2001 Jan-Mar;64(1):15-9. PMID 11322061
- [Background] Singh V, Kumar B, Nain CK, Singh B, Sharma N, Bhalla A, Sharma AK. Noradrenaline and albumin in paracentesis-induced circulatory dysfunction in cirrhosis: a randomized pilot study. J Intern Med. 2006 Jul;260(1):62-8. doi: 10.1111/j.1365-2796.2006.01654.x. PMID 16789980
- [Background] Appenrodt B, Wolf A, Grunhage F, Trebicka J, Schepke M, Rabe C, Lammert F, Sauerbruch T, Heller J. Prevention of paracentesis-induced circulatory dysfunction: midodrine vs albumin. A randomized pilot study. Liver Int. 2008 Aug;28(7):1019-25. doi: 10.1111/j.1478-3231.2008.01734.x. Epub 2008 Apr 11. PMID 18410283
- [Background] Sanyal AJ, Boyer T, Garcia-Tsao G, Regenstein F, Rossaro L, Appenrodt B, Blei A, Gulberg V, Sigal S, Teuber P; Terlipressin Study Group. A randomized, prospective, double-blind, placebo-controlled trial of terlipressin for type 1 hepatorenal syndrome. Gastroenterology. 2008 May;134(5):1360-8. doi: 10.1053/j.gastro.2008.02.014. Epub 2008 Feb 13. PMID 18471513
- [Background] Martin-Llahi M, Pepin MN, Guevara M, Diaz F, Torre A, Monescillo A, Soriano G, Terra C, Fabrega E, Arroyo V, Rodes J, Gines P; TAHRS Investigators. Terlipressin and albumin vs albumin in patients with cirrhosis and hepatorenal syndrome: a randomized study. Gastroenterology. 2008 May;134(5):1352-9. doi: 10.1053/j.gastro.2008.02.024. Epub 2008 Feb 14. PMID 18471512
- [Background] Gadano A, Moreau R, Vachiery F, Soupison T, Yang S, Cailmail S, Sogni P, Hadengue A, Durand F, Valla D, Lebrec D. Natriuretic response to the combination of atrial natriuretic peptide and terlipressin in patients with cirrhosis and refractory ascites. J Hepatol. 1997 Jun;26(6):1229-34. doi: 10.1016/s0168-8278(97)80456-4. PMID 9210608
- [Background] Valla D, Lee SS, Moreau R, Hadengue A, Sayegh R, Lebrec D. [Effects of glypressin on the splanchnic and systemic circulation in patients with cirrhosis]. Gastroenterol Clin Biol. 1985 Dec;9(12):877-80. French. PMID 3830801
- [Background] Arroyo V, Gines P, Gerbes AL, Dudley FJ, Gentilini P, Laffi G, Reynolds TB, Ring-Larsen H, Scholmerich J. Definition and diagnostic criteria of refractory ascites and hepatorenal syndrome in cirrhosis. International Ascites Club. Hepatology. 1996 Jan;23(1):164-76. doi: 10.1002/hep.510230122. No abstract available. PMID 8550036